CLINICAL TRIAL: NCT01720797
Title: Alveolar Microperforation for Inflammation-Enhanced Tooth Movement During Orthodontic Treatment
Acronym: Propel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: AlevoLogic LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20121593
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Malocclusion
Keywords: Malocclusion; Accelerated tooth movement; Braces; Orthodontic treatment; Propel
MeSH Terms: conditions — Malocclusion | interventions — Anesthetics, Local; Chlorhexidine; chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Micro-osteoperforation (Experimental): Minimally invasive micro-osteoperforation (PROPEL™) procedure used to achieve rapid orthodontic tooth movement. Topical or local anesthetic will be delivered in the area to be treated in accordance with standard practice. Prior to intervention subject will swish 5cc of chlorhexidine for one minute, twice, will take place. Following procedure Chlorhexidine rinses are to begin twice a day for a week.
  Interventions: Device: Micro-osteoperforation; Drug: Anesthestic; Other: Chlorhexidine
- Non Micro-osteoperforation (Other): Prior to intervention a swish of 5cc of chlorhexidine for one minute, twice, will take place. Chlorhexidine rinses are to begin twice a day for a week.
  Interventions: Other: Chlorhexidine

INTERVENTIONS:
Device: Micro-osteoperforation — Minimally invasive micro-osteoperforation procedure used to achieve rapid orthodontic tooth movement.
  Other Names: PROPEL™
  Arms: Micro-osteoperforation
Drug: Anesthestic — Topical or local anesthetic will be delivered in the area to be treated in accordance with standard practice.
  Other Names: Topical or local anesthetic
  Arms: Micro-osteoperforation
Other: Chlorhexidine — Prior to intervention subject will swish 5cc of chlorhexidine for one minute, twice. Following procedure Chlorhexidine rinses are to begin twice a day for a week.
  Other Names: Peridex

SUMMARY:
The purpose of this research study is to assess the clinical effectiveness of the procedure of a minimally invasive alveolar microperforation procedure to achieve accelerated tooth movement in patients undergoing orthodontic treatment. "Accelerated tooth movement" means that using the PROPEL™ device may help complete your treatment with braces on one side of your mouth sooner than would be expected if the device were not to be used.

DETAILED DESCRIPTION:
Following informed consent and satisfying the screening/enrollment assessments, a panoramic and periapical radiograph of the teeth designated for micro-osteoperforation treatment is to be taken. Prior to the intervention the subjects will swish 5cc of chlorhexidine for one minute, twice. Micro-osteoperforation, PROPEL™, is conducted under local or topical anesthesia AFTER the subject is banded and bonded. The procedure will be randomized to either the left or right side in each subject. Following the procedure, Chlorhexidine rinses are to begin twice a day for a week.

The subjects will be advised to take Tylenol only in case of significant pain. Subjects will be seen four to six weeks after completion of treatment for the first follow-up. Subjects will be followed up with a telephone consult 24 hours after micro-osteoperforation is performed. They will be asked if any pain medication was taken after being dismissed from the research center and if so, they will be asked the name and dose of medication taken.

Study will conclude at the 6 month follow up visit or when space on the treating side is closed.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent and adult subjects ages 18-55 years old, in good general health, with adult or mixed dentition, regardless of presence of third molars.
* Subjects are American Society of Anesthesiologists (ASA) class I (ASA class I - Patients are considered to be normal and healthy).
* Periodontal or gingivitis diseases must be addressed prior to study enrollments: Probing Depth(PD)<5mm,Gingival Index (GI)<1,Plaque Index(PI)=1
* If any caries is present, patient will be referred to dentist for treatment and maintenance before beginning treatment
* Able to understand English, follow simple instructions and sign informed consent

Exclusion Criteria:

* Subjects who have taken any local or systemic antibiotics, corticosteroids or periodontal medications in the previous six weeks.
* Subjects with extreme skeletal class II malocclusion: Overjet>10mm, (Pogonion to Nasion Perpendicular line)Pg-Nper>18mm, A point Nasion B point (ANB)>7, Sella Nasion line to Gonion Gnathion Line (SN-GoGN)>38
* Vulnerable subjects who unable to consent for themselves

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Calogero Dolce, D.D.S, PhD, Principal Investigator — University of Florida, Interim Chair
Locations (1):
- University of Florida, Department of Orthodontics, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Micro-osteoperforation: Minimally invasive micro-osteoperforation procedure used to achieve rapid orthodontic tooth movement. Topical or local anesthetic will be delivered in the area to be treated in accordance with standard practice. Prior to intervention subject will swish 5cc of chlorhexidine for one minute, twice, will take place. Following procedure Chlorhexidine rinses are to begin twice a day for a week.
  Micro-osteoperforation: Minimally invasive micro-osteoperforation procedure used to achieve rapid orthodontic tooth movement.
  Anesthestic: Topical or local anesthetic will be delivered in the area to be treated in accordance with standard practice.
  Chlorhexidine: Prior to intervention subject will swish 5cc of chlorhexidine for one minute, twice. Following procedure Chlorhexidine rinses are to begin twice a day for a week.
Period: Overall Study
Arm/Group | Micro-osteoperforation | Non Micro-osteoperforation
Started | 12 | 9
Completed | 9 | 9
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Micro-osteoperforation: Minimally invasive micro-osteoperforation procedure used to achieve rapid orthodontic tooth movement. Topical or local anesthetic will be delivered in the area to be treated in accordance with standard practice. Prior to intervention subject will swish 5cc of chlorhexidine for one minute, twice, will take place. Following procedure Chlorhexidine rinses are to begin twice a day for a week.
- Total: Total of all reporting groups
Arm/Group | Micro-osteoperforation | Non Micro-osteoperforation | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 9 | 21
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Tooth Movement Between the Groups
Description: Accelerated tooth movement effectiveness as measured by dental impressions. These impressions at the 6 month follow-up will evaluate the rate of tooth movement by measuring casts.
  Ortholnsight software was used to measure the millimeters of tooth movement from the dental impressions, and then was converted to a Mean and Standard Deviation measurement.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of movement
Arm/Group | Micro-osteoperforation | Non Micro-osteoperforation
Number analyzed (Participants) | 9 | 9
percentage of movement | 4.345 (1.257) | 4.04 (0.991)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Micro-osteoperforation | Non Micro-osteoperforation
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No